CLINICAL TRIAL: NCT04948294
Title: Comparison of the Intubation Condition Between Using Two Types of Blade in Patients Receiving Tracheal Intubation Using Videolaryngoscope: Channeled Blade vs. Non-channeled Blade
Brief Title: Comparison of the Intubation Condition Between Two Different Types of Video Laryngoscope Blades
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Hyungseok Seo, Assistant Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KHNMC 2019-07-020-001
Record Dates: First submitted 2021-06-26; First posted 2021-07-01 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Intubation Complication

STUDY DESIGN:
Intervention Model Description: Patients requiring tracheal intubation for general anesthesia
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Channeled group (Experimental): Group of patients using a channeled blade for videolaryngoscopy
  Interventions: Device: Channeled blade
- Non-channeled group (Active Comparator): Group of patients using a non-channeled blade (standard type) for videolaryngoscopy
  Interventions: Device: Non-channeled blade

INTERVENTIONS:
Device: Channeled blade — In the present group, a tracheal tube was launched in the channel of the blade before tracheal intubation
  Arms: Channeled group
Device: Non-channeled blade — In the present group, a tracheal tube was not launched in the videolaryngoscope blade before tracheal intubation
  Arms: Non-channeled group

SUMMARY:
The present study compares two different types of videolaryngoscope blade, which is a channeled and non-channeled blade. The purpose of the study is to investigate the effect of the type of videolaryngoscope blade on the intubation condition.

DETAILED DESCRIPTION:
In tracheal intubation for general anesthesia, one of the two types of the blade during a video laryngoscopy can be used, one is a channeled blade that has a channel for tracheal tube launching, the other is a non-channeled blade. In the present study, the outcomes by using two types of the videolaryngoscope blade such as the intubation condition, intubation time, first-pass rate, and the incidence of intubation-related complications were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving tracheal intubation for general anesthesia
* Patients with physical status 1, 2, or 3 by American Society of Anesthesiologists Physical Status.

Exclusion Criteria:

* Body mass index <18.5 kg/m2 or >35 kg/m2
* Patients with a history of airway surgery
* Patients with increased risk of aspiration
* Patients who have any pathology (polyp, tumor, or inflammation) in the upper airway and larynx

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Intubation time | Immediately after tracheal intubation completed
  the time for tracheal intubation

SECONDARY OUTCOMES:
First-pass rate | Immediately after tracheal intubation completed
  the success rate of tracheal intubation with one attempt
Intubation-related complications | within 24 hours after surgery
  the incidence of overall complications related with tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Hyungseok Seo, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Gangdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No